CLINICAL TRIAL: NCT02048579
Title: Increasing Academic Success in Middle School Students With ADHD
Acronym: STAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R34MH092466-01A1 (NIH)
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Behavior Therapy + MI Intervention (Supporting Teens' Academic Needs Daily); Treatment as Usual
MeSH Terms: interventions — Behavior Therapy; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (No Intervention)
- Behavior Therap + Motivational Interviewing (Experimental): Supporting Teens' Academic Needs Daily Therapy program delivered to parents and teens
  Interventions: Behavioral: Behavior Therapy + Motivational Interviewing

INTERVENTIONS:
Behavioral: Behavior Therapy + Motivational Interviewing
  Other Names: Supporting Teens' Academic Needs Daily (STAND)
  Arms: Behavior Therap + Motivational Interviewing

SUMMARY:
Broadly, the purpose of the proposed study is to test the efficacy of a parent-coordinated, parent-teen-teacher collaborative intervention for middle school students with ADHD and academic impairment (STAND; Supporting Teens' Academic Needs Daily). [This model was chosen because of its potential ability to promote treatment maintenance and generalizability across school years, because parents will be taught to implement, monitor, and adjust intervention components as needed. Key innovative components in the STAND intervention address previously reported treatment barriers: 1) a parent-delivered academic intervention to promote maintenance and generalization across school years, and to relieve some of the burden of intervention delivery from teachers, 2) motivational interviewing to address parent disengagement from and adolescent resistance to the treatment process, 3) multiple tailored options for home-school communication, including a web-based support system, to facilitate home-school communication, and 4) empowering parents by coaching them to effectively and tactfully involve teachers in the treatment planning and monitoring process in order to increase teachers' willingness to support the child's academic needs. To study the feasibility and preliminary efficacy of the STAND treatment model,] two cohorts of 42 middle school students with ADHD will be recruited (total N=84) and randomly assigned to participate in STAND or a treatment-as-usual monitoring group. All participants will complete intake, mid-treatment, post-treatment, [and follow-up] assessments designed to monitor academic functioning, [intervention feasibility, compliance, and satisfaction].

Aim 1: The proposed study will evaluate the efficacy, [maintenance, and cross-school year generalization] of a parent-teen-teacher collaborative intervention (Supporting Teens' Academic Needs Daily; STAND) vs. treatment as usual to increase the academic functioning of middle school students with ADHD. Intervention effects on ADHD symptomatology and impairment, grade-point-average (GPA), [organization, daily planner use], homework completion, teacher ratings of academic functioning and classroom behavior, and the parent-teen relationship will be examined.

Aim 2: The proposed study will examine the acceptability and feasibility of the STAND program. Parents and teens will report on [satisfaction, barriers to treatment participation, therapeutic alliance, and treatment credibility] throughout the intervention and follow-up period. [Therapists will also complete ratings of parent and adolescent engagement and compliance with treatment procedures] will be collected from participants in the program. Parent, teen, and teacher compliance with intervention procedures will also be measured in order to assess feasibility. Treatment fidelity measures will also be collected in order to measure clinician adherence to the manualized STAND procedures.

Aim 3: The proposed study will also explore ways to improve home-school communication during the middle school years. To this end, families will be given options regarding the modality of communication with teachers, and parent, teen, and teacher preferences for medium of intervention delivery will be examined (i.e., web-based, email, paper/pencil).

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR ADHD Diagnosis; regular education placement in school; academic impairment

Exclusion Criteria:

* IQ<80; Autism or PDD diagnosis;

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2012-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Grade Point Average | One year

SECONDARY OUTCOMES:
Parent Rated Adolescent Academic Problems | One Year
parent rated ADHD symptoms | one year

CONTACTS AND LOCATIONS:
Overall Officials: Margaret H Sibley, Ph.D., Principal Investigator — Florida International University; Willam Pelham, Ph.D., Principal Investigator — Florida International University